CLINICAL TRIAL: NCT01105819
Title: A Study Comparing a Suspension of Lactobacillus Plantarum 299 With Chlorhexidine for Oral Care in Intubated Mechanically Ventilated Patients in Intensive Care
Brief Title: Chlorhexidine vs Lactobacillus Plantarum for Oral Care in Intubated ICU Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: County Council of Halland, Sweden (Other Government); Probi AB (Industry)
Responsible Party: Principal Investigator, Bengt Klarin, Consultant, MD, PhD, Region Skane
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PROHYG 1B
Record Dates: First submitted 2010-04-09; First posted 2010-04-19 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Pathogenic Bacteria in the Oropharynx; Ventilator-associated Pneumonia
Keywords: Probiotics; Lactobacillus plantarum 299; Ventilator-associated pneumonia VAP; Chlorhexidine; Tracheal secretions; Oropharyngeal secretions
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Chlorhexidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard oral care with chlorhexidine (Other): The control group will receive a standard oral care. This includes suction of secretions, brushing of teeth cleansing of the oral cavity with swabs soaked with a chlorhexidine solution. This procedure is performed twice a day. In between, suction whenever needed and cleansing with swabs soaked with carbonated bottled water is performed
  Interventions: Procedure: Chlorhexidine for standard oral care
- Lactobacillus plantarum 299 (Active Comparator): The study group will be attended in the same manor but the swabs used for cleansing are soaked with carbonated water directly from freshly opened bottles. As the final part of the procedure oral mucosal surfaces are pencilled with a suspension of the probiotic bacterium Lactobacillus plantarum 299 Cultures from the oropharynx and tracheal secretions are taken at inclusion (day 1) and then on days 2,3,5,7,10,14 and 21 or before extubation if this occurs on a non-culture day
  Interventions: Procedure: Lactobacillus plantarum 299 for oral care

INTERVENTIONS:
Procedure: Lactobacillus plantarum 299 for oral care — The study group will be attended in the same manor but the swabs used for cleansing are soaked with carbonated water directly from freshly opened bottles. As the final part of the procedure oral mucosal surfaces are pencilled with a suspension of the probiotic bacterium Lactobacillus plantarum 299 Cultures from the oropharynx and tracheal secretions are taken at inclusion (day 1) and then on days 2,3,5,7,10,14 and 21 or before extubation if this occurs on a non-culture day
  Arms: Lactobacillus plantarum 299
Procedure: Chlorhexidine for standard oral care — A The control group will receive the standard oral care of the department (general ICU, Lund University Hospital).
  This includes suction of secretions, brushing of teeth cleansing of the oral cavity with swabs soaked with a chlorhexidine solution. This procedure is performed twice a day. In between, suction whenever needed and cleansing with swabs soaked with carbonated bottled water is performed Cultures from the oropharynx and tracheal secretions are taken at inclusion (day 1) and then on days 2,3,5,7,10,14 and 21 or before extubation if this occurs on a non-culture day
  Arms: Standard oral care with chlorhexidine

SUMMARY:
Critically ill patients often need ventilatory support through a plastic tube connected to a ventilator. Those patients have a altered microbiological flora in the mouth, oropharynx as well as throughout the intestine. Bacteria that can cause illness are often found in the oropharynx in such patients and measures are taken in order to reduce the risk of secondary infections by those bacteria. In all intensive care patients oral care is provided by the nursing staff aiming at a reduction of the pathogenic species. This is done by a variety measures.

Chlorhexidine (CHX) is an antisepticum with a capability to reduce bacterial counts in the mouth and oropharynx and has been shown to be of value also for intubated patients. It is used frequently throughout the world.

Ventilator-associated pneumonia (VAP) is a costly rather frequent complication to intensive care and mechanical ventilation and is usually caused by aspiration of infected secretions from the oropharynx. CHX has in some studies been shown to reduce the frequency of VAP.

The probiotic bacterium Lactobacillus plantarum 299 has the ability to adhere to the mucosa throughout the gastro-intestinal tract including the mouth and in our pilot study we found that L plantarum had better ability to reduce colonisation with enteric bacteria in the oropharynx than CHX had. Figures not statistical significant so this present study is aiming to get a larger amount of data.

The procedure was found to be safe Hypothesis: Lactobacillus plantarum is better than CHX for the reduction of pathogenic bacteria in the oropharynx in intubated mechanically ventilated patients and consequently has a better potential to reduce the frequency of VAP

DETAILED DESCRIPTION:
This study is an expansion of a pilot study performed at the ICU Lund University Hospital, Sweden where 50 patients were included (ISRCTN00472141).

Results have been published in Critical Care 2008, 12:R136 The protocol is the same and in this second phase we intend to include 100 patients and results will be summed up.

Three centres are engaged. The results from the pilot study is encouraging and we are aiming at getting statistical significance in the differences in pathogenic findings in the cultures from oropharynx and also better a better basis for the calculation of the number of patients needed to get sufficient power to study difference in VAP frequency.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Critically ill patients anticipated to require mechanical ventilation for at least 24 hours

Exclusion Criteria:

* Pneumonia as admission diagnosis,
* Fractures on the facial skeleton or the skull base;
* Known ulcers in the oral cavity, the oropharynx, or the esophagus
* Known immune difficency
* Carrier of HIV or Hepatitis
* Patient being moribund

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-04; Primary Completion 2016-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
To compare the number and frequency of cultures with pathogenic bacteria and fungi from the oropharynx and tracheal secretions and the spectra of these microbiological species | During study time in connection with the care in the ICU until invasive mechanical ventilation is terminated
Recovery of Lactobacillus plantarum 299 in tracheal secretions in the active treatment group as an indicator of aspiration | During study time in connection with the care in the ICU until invasive mechanical ventilation is terminated

SECONDARY OUTCOMES:
SOFA score and Influence on lung function measured as Lung Injury Severity Score | From admission to the ICU til discharge from the ICU
Difference in emerge of Ventilator Associated Pneumonia | During ICU stay
Validation of micobiological findings compared to the use of antibiotics | ICU stay + 48 hours
C-reactive protein and white blood cell counts | From admission to the ICU til discharge from the ICU
Evaluation of microbiological cultures taken on clinical grounds | ICU-stay + 48 hours
  We want to examine the possible influence of the added probioticum on the frequence of positive cultures from other sites than those taken per protocol.
  Samples taken during ICU-stay and 48 hours after discharge from the ICU will be examened The type of species in positive cultures are also of interest. Blood cultures may act as indicator of vascular spread of the studied bacterium.
  According to the protocol samples for blood cultures are not taken
28 day mortality | 28 days after ICU admission
6 months mortality | 6 months after ICU admission

CONTACTS AND LOCATIONS:
Locations (3):
- Sweden (3):
  - Intensive Care Unit, Halmstad Central Hospital, Halmstad
  - Intensive Care Unit, Kristianstad Central hospital, Kristianstad
  - Intensive Care Unit, Lund University Hospital, Lund

IPD SHARING:
Plan to Share IPD: Yes
Results are under review and are planned for publishing in a scientific journal

REFERENCES:
- [Result] Klarin B, Molin G, Jeppsson B, Larsson A. Use of the probiotic Lactobacillus plantarum 299 to reduce pathogenic bacteria in the oropharynx of intubated patients: a randomised controlled open pilot study. Crit Care. 2008;12(6):R136. doi: 10.1186/cc7109. Epub 2008 Nov 6. PMID 18990201
- [Derived] Klarin B, Adolfsson A, Torstensson A, Larsson A. Can probiotics be an alternative to chlorhexidine for oral care in the mechanically ventilated patient? A multicentre, prospective, randomised controlled open trial. Crit Care. 2018 Oct 28;22(1):272. doi: 10.1186/s13054-018-2209-4. PMID 30368249